CLINICAL TRIAL: NCT03056963
Title: Guided Imagery Training and Self-Referential Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTEXAS-2016-07-0080
Record Dates: First submitted 2017-02-10; First posted 2017-02-17 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Depression; Negative Thoughts
Keywords: Guided Imagery
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Self-Reference Training (Experimental): Participants in this arm will complete the Positive Self-Reference Training (PSRT).
  Interventions: Behavioral: Positive Self-Reference Training
- Neutral Training Control (Placebo Comparator): Participants in this arm will complete the neutral training paradigm.
  Interventions: Behavioral: Neutral Training Control

INTERVENTIONS:
Behavioral: Positive Self-Reference Training — Participants in this intervention will review a brief psychoeducational video describing the training, and then be given cues every other day designed to practice skills. Participants will then practice visualizing and describing scenes based on these cues. This training will be focused on positive self-referent material.
  Arms: Positive Self-Reference Training
Behavioral: Neutral Training Control — Participants in this intervention will review a brief psychoeducational video describing the training, and then be given cues every other day designed to practice skills. Participants will then practice visualizing and describing scenes based on these cues. This training will be focused on neutral, non-self-referent material.
  Arms: Neutral Training Control

SUMMARY:
The purpose of this study is to examine the efficacy of a guided imagery paradigm for reducing negative ways of thinking about the self. There will be at least 60 participants enrolled at the University of Texas at Austin. Participants will be randomly selected to receive one of two types of trainings, each over the course of two weeks. Participants will undergo the training exercises at home. The training exercises will help them to think differently about themselves.

Participants will be able to determine if they are eligible, and then participate, by filling out a screening questionnaire online.

DETAILED DESCRIPTION:
This study uses a randomized controlled trial to compare two types of guided imagery. One intervention is an active intervention; the other is intended to be inert. These interventions were developed based on extensive research indicating the efficacy of using imagery in depression, and a perceived lack of treatments targeting biased self-referential processing.

This protocol aims to develop a novel intervention which can be used on its own or as an adjunct to existing treatments. Common treatments for Major Depressive Disorder (MDD) are diffuse; this paradigm instead aims to specifically target negative self-schema, a part of the cognitive model of MDD. This study focuses on participants with elevated depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to provide informed consent
* elevated depressive symptoms -- i.e., a score above a 13 on the Center for Epidemiologic Studies Depression Scale (CESD)

Exclusion Criteria:

* N/A

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Change in response on the Self-Referent Encoding Task (SRET) | Participants will complete the SRET at baseline, after one week, and after two weeks. Change will be assessed primarily as SRET at two weeks MINUS SRET at baseline.
  The SRET is a task that asks participants to categorize words as self-referential or not. Its outcomes are focused on behavioral response and reaction time. We have shown that it has good test-retest reliability over the course of one week.

SECONDARY OUTCOMES:
Depressive Symptomatology | Participants will complete measures of depressive symptoms at baseline, after one week, and after two weeks.
  Measures of depressive symptoms will be measured with the CESD, a self-report questionnaire used in the literature to measure levels of depression. This questionnaire has good test-retest reliability, and reliably changes with symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Dainer-Best, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Screening Questionnaire — https://redcap.prc.utexas.edu/redcap/surveys/?s=DCXW77HAF3